CLINICAL TRIAL: NCT00133705
Title: Randomized Control Trial Of Mifepristone for Fibroids
Brief Title: Trial of Mifepristone for Fibroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kevin Fiscella, Tenured Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RO1-HD042578-2; R01HD042578 (NIH)
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Results first posted 2012-11-30 (Estimated); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Leiomyoma
Keywords: A benign tumor derived from smooth uterine muscle tissue.
MeSH Terms: conditions — Leiomyoma | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mifepristone (Experimental): Mifepristone 5 MG capsule taken once daily by mouth
  Interventions: Drug: Mifepristone
- Inert capsule (Placebo Comparator): Placebo (for Mifepristone) capsule of nearly identical color, size, and weight taken once daily by mouth
  Interventions: Drug: Inert Capsule

INTERVENTIONS:
Drug: Mifepristone — Mifepristone 5mg/day by mouth for 6 months
  Other Names: RU486
  Arms: Mifepristone
Drug: Inert Capsule — sugar pill
  Arms: Inert capsule

SUMMARY:
The purpose of this trial is to determine if low-dose mifepristone benefits women with symptomatic fibroids.

DETAILED DESCRIPTION:
This trial is designed to assess the efficacy and tolerability of mifepristone 5 mg given daily for 6 months to pre-menopausal women with symptomatic fibroids. The primary study outcome will be disease-specific quality of life. Secondary outcome measures include global quality of life, pain, bleeding, potential adverse effects, tumor size, and endometrial effects. The researchers will also examine a the effect of mifepristone on uterine blood flow. Randomization of study subjects will be stratified in order to ensure that equal numbers of women with moderate and severe symptoms will be enrolled in the placebo and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Female
* Age: 18 - premenopausal
* Have at least moderate symptoms of menorrhagia or pelvic pain/pressure
* Have a total uterine volume greater than or equal to 160 cc by ultrasound measurement and at least one fibroid that is => 2.5cm in size
* Have a score of equal to or greater than 39 on the Uterine Fibroid Symptom and Quality of Life scale
* Declined standard treatment options for symptomatic fibroids
* Agree to use a double-barrier method (condoms, diaphragms) or other effective non-hormonal methods of contraception (abstinence, sterilization) throughout participation in the study to prevent pregnancy and to report any exposure to pregnancy to the research staff immediately
* Willing and able to give informed consent
* Willing and able to comply with study requirements

Exclusion Criteria:

* Current or planned pregnancy during the study period
* Menopausal, as indicated by follicle stimulating hormone (FSH) level of the reference laboratory
* Currently breast-feeding
* Untreated abnormal pap smear
* Presence of conditions other than fibroids contributing to pain and/or bleeding
* Hemoglobin < 9.0 mg/dl
* Presence of adnexal masses or tenderness indicating further evaluation or surgery
* Grade III or IV hydronephrosis by ultrasound
* Severe, active mental health disorder
* Active substance abuse or dependence
* Presence of any contraindication to mifepristone including:

  * Adrenal insufficiency by history
  * Sickle cell disease
  * Active liver disease (liver function tests greater than 1.5 times upper range of normal)
  * Severe, respiratory disease (P02 saturation< 92%)
  * Renal disease (serum creatinine > 1.5 mg/dl)
  * Blood clotting defect. (abnormal PT and PTT)
  * Thromboembolic disease (history of deep vein thrombosis or pulmonary embolus)
* Current or recent (within the past 3 months) use of the following medications:

  * Oral or systemic corticosteroids
  * Hormones: estrogens, progestins, oral contraceptives
  * Danazol, anticoagulants
* Herbal or botanical supplements with possible hormonal effects.
* Use within the past six months of the gonadotropin releasing hormones (GnRH) analogs or Depo-Provera.
* Current or planned use during the study of any of the following medications/or products:

  * ketoconazole,
  * itraconazole,
  * erythromycin,
  * grapefruit juice,
  * rifampin,
  * St John's Wort,
  * phenytoin,
  * phenobarbital, or
  * carbamazepine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2003-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Fiscella, MD, MPH, Principal Investigator — University of Rochester School of Medicine & Dentistry
Locations (1):
- University of Rochester School of Medicine & Dentistry, Rochester, New York, United States

REFERENCES:
- [Background] Eisinger SH, Bonfiglio T, Fiscella K, Meldrum S, Guzick DS. Twelve-month safety and efficacy of low-dose mifepristone for uterine myomas. J Minim Invasive Gynecol. 2005 May-Jun;12(3):227-33. doi: 10.1016/j.jmig.2005.01.022. PMID 15922980
- [Background] Eisinger SH, Meldrum S, Fiscella K, le Roux HD, Guzick DS. Low-dose mifepristone for uterine leiomyomata. Obstet Gynecol. 2003 Feb;101(2):243-50. doi: 10.1016/s0029-7844(02)02511-5. PMID 12576246
- [Derived] Fiscella K, Eisinger SH, Meldrum S, Feng C, Fisher SG, Guzick DS. Effect of mifepristone for symptomatic leiomyomata on quality of life and uterine size: a randomized controlled trial. Obstet Gynecol. 2006 Dec;108(6):1381-7. doi: 10.1097/01.AOG.0000243776.23391.7b. PMID 17138770

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were recruited between March 3, 2004 and March 30, 2005 through local media and contacts with community physicians.
Pre-assignment Details: 38 women were deemed ineligible. Of those exclusion criteria applied to 27 and 11 declined participation.
Groups:
- Treatment Group: This group will receive 5 mg. capsules to be taken once daily.
- Placebo Group: These women received placebo capsules identical in appearance and weight to the 5 mg. mifepristone capsule to be taken once daily.
Period: Overall Study
Arm/Group | Treatment Group | Placebo Group
Started | 22 | 20
Completed | 20 | 17
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Mifepristone 5 mg.: Twenty-two women received 5 mg. mifepristone daily.
- Placebo: Twenty women received a placebo pill daily.
- Total: Total of all reporting groups
Arm/Group | Mifepristone 5 mg. | Placebo | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 20 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (6.2) | 43.2 (4.7) | 43.0 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Uterine Volume
Description: Uterine volume is measured in mLs
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 22 | 20
mL | 719 (663) | 449 (236)

ADVERSE EVENTS:
Arm/Group | Treatment Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/20

LIMITATIONS AND CAVEATS:
There were no adverse events in this clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No